CLINICAL TRIAL: NCT02437682
Title: Translation and Validation of the PASS Test for Gastro-esophageal Reflux Disease (GERD) Patients With Partial Response to PPI in Chinese Population: PASS-HK
Brief Title: Translation and Validation of the PASS Test for GERD Patients With Partial Response to PPI: PASS-HK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justin Che-Yuen Wu, Professor, Chinese University of Hong Kong
Other Study IDs: PASS-HK
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Gastro-esophageal Reflux Disease
Keywords: Gastro-esophageal Reflux Disease; Proton pump inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PASS test is only available and valid tool for the evaluation of persistent acid-related symptoms in patients receiving PPI therapy. There is lack of a validated Chines version of PASS questionnaire for the GERD patients with partial response to proton pump inhibitor (PPI). The English version of PASS test will be translated to traditional Chinese by using forward-backward procedure, and the Chinese version of PASS test will be validated its psychometric properties in Hong Kong population.

Eligible subjects will be invited to administer questionnaires to evaluate the psychometric properties of the Chinese version of PASS test.

DETAILED DESCRIPTION:
Gastro-esophageal reflux disease (GERD) is a common condition defined as symptoms or mucosal damage produced by the abnormal reflux of gastric contents into the esophagus. Symptoms highly specific for GERD are heartburn, regurgitation, or both, which often occur after meals. The prevalence of GERD is around 20% for weekly reflux symptoms in the Western population, while 9.3% in Chinese population. However, approximately 20-30% of patients with GERD experience only a partial response of their heartburn of regurgitation symptoms to PPI therapy.

There is lack of a validated Chines version of PASS questionnaire for the GERD patients with partial response to PPI.

Before a treatment response assessment tool can be used clinically, various questions on reliability and validity of the instrument need to be addressed. The aims of this study are (1) to translate the PASS test from English to traditional Chinese, named PASS-HK, and (2) to assess the psychometric properties of the PASS-HK, before clinical application.

Linguistic translation of the PASS questionnaire from English to Chinese version will follow a forward-backward procedure.

After finalization of Chinese version of the PASS (PASS-HK), the reliability of PASS-HK will be evaluated for internal consistency using Cronbach's alpha. The intraclass correlation coefficient was calculated within 14 days for two surveys in order to evaluate the reproducibility of the results under constant conditions. Pearson product moment correlation coefficient will be used to evaluate whether PASS-HK can measure what it claims to measure by comparing with SF-12v2, GERD QOL and GREDSQ scores.

All eligible subjects will be invited to complete PASS-HK twice within 14 days under a stable condition. In addition to PASS-HK, all patients will have to complete SF-12v2, GERD-QOL, GERDQ and GERDSQ questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Able to give study informed consent
* Male or female. Age 18 or above
* Have at least 6 months history of GERD symptoms (need not to be consecutive) as chief complaint, e.g. acid regurgitation or heartburn
* Subject has been taking any PPI at standard dose for at least 8 weeks Subject has persistent symptoms during PPI therapy with GERDQ score ≥8
* An upper gastrointestinal endoscopy is required within the past 1 year to confirm the absence of mucosal breaks, peptic ulcer and other GI diseases e.g. gastric outlet obstruction

Exclusion Criteria:

* Patients that have not experienced any GERD symptom improvement at all during PPI treatment
* Unstable or clinically significant cardiovascular, respiratory, hepatic, renal, metabolic, psychiatric, other clinical disorders, or gastrointestinal and esophageal disorders besides GERD. Clinically significant is defined as disorders that could compromise patients' safety or interfere with the evaluation of the study as judged by the investigator.
* History of or current malignant disease
* Subject is pregnant or lactating
* Prior surgery of the upper GI tract (open, endoscopic and laparoscopic surgery on the esophagus, the stomach and the duodenum)
* Illiterate patient (who cannot administer questionnaire)
* Known hypersensitivity to any PPI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject has been taking any PPI and still has persistent GERD symptoms during PPI therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
PASS_C questionnaire | One year
  the reliability of PASS-HK will be evaluated for internal consistency using Cronbach's alpha. The intraclass correlation coefficient will be calculated within 14 days for two surveys in order to evaluate the reproducibility of the results under constant conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Justin C.Y. Wu, MBChB(CUHK), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No